CLINICAL TRIAL: NCT02082548
Title: An International Multicenter Clustered Randomized Controlled Trial to imProve Treatment With AntiCoagulanTs in Patients With Atrial Fibrillation.
Brief Title: Clinical Trial to Improve Treatment With Blood Thinners in Patients With Atrial Fibrillation
Acronym: IMPACT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Daiichi Sankyo (Industry); Boehringer Ingelheim (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00049709
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; anticoagulation; education; educational intervention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): educational intervention arm
  Interventions: Other: Educational Intervention
- control (No Intervention): Standard of care

INTERVENTIONS:
Other: Educational Intervention — This intervention will contain educational materials for both patients and providers that are specific to the needs in each participating country
  Arms: Intervention

SUMMARY:
To determine whether a comprehensive evaluation and customized multilevel educational interventions will increase the rate of use of oral anticoagulants and the adherence and persistence of use in patients with atrial fibrillation. Our hypothesis is that there will be differences in the use of oral anticoagulants and the persistence in patients between the control and interventional group. There will be a greater change in the use of oral anticoagulants over one year in the cohort in the intervention sites than the control sites. This will be due to two factors: greater initiation of oral anticoagulants among patients not treated at baseline and greater persistence of treatment for those on treatment at baseline

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients over the age of 18 with paroxysmal, persistent or permanent atrial fibrillation who have a 12-lead ECG showing atrial fibrillation and/or more than one rhythm strip showing atrial fibrillation at least 2 weeks apart, not due to a reversible cause (like post-CABG))
* 2. At least one of the traditional CHADS2 risk factors or at least two CHA2DS2 VASc risk factors

Exclusion Criteria:

* Mechanical prosthetic valve
* Clinically unstable at the time of enrollment (ie, with ongoing shock)
* Terminal illness and/or comfort care
* Unable to provide consent (e.g. severe cognitive impairment)
* Patients unable to have one year of follow-up for any reason
* Clear and absolute contraindication to oral anticoagulation (for example, active bleeding or recent life-threatening bleeding such as ICH)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2374 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Change in proportion of patients taking oral anticoagulants | 1 year
  Change in proportion of patients taking oral anticoagulants from baseline to one year

SECONDARY OUTCOMES:
Change in proportion of patients able to continue anticoagulation | 1 year
  Change in proportion of patients able to continue anticoagulation for one year
Change in proportion of patients who are not on anticoagulation at baseline and are on anticoagulation | 1 year
  Change in proportion of patients who are not on anticoagulation at baseline and are on anticoagulation at one year
Death, total | 1 year
Stroke, hemorrhagic and non-hemorrhagic | 1 year
Major and non-major clinically relevant bleeding | 1 year

OTHER OUTCOMES:
Systemic Embolism | 1 year
Transient Ischemic Attack | 1 year
Hospitalizations for cardiovascular causes | 1 year
Time in therapeutic range for patients on vitamin K antagonists (VKA) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Granger, MD, Principal Investigator — Duke Clinical Research Institute
Locations (5):
- INECO Neurosciencias Orono, Rosario, Santa Fe Province, Argentina
- Federal University of Sao Paulo, São Paulo, Brazil
- Peking University First Hospital, Beijing, China
- St Johns Medical College, Bangalore, India
- University of Medicina and Pharmacy Carol Davila, Bucharest, Romania

REFERENCES:
- [Derived] Vinereanu D, Lopes RD, Bahit MC, Xavier D, Jiang J, Al-Khalidi HR, He W, Xian Y, Ciobanu AO, Kamath DY, Fox KA, Rao MP, Pokorney SD, Berwanger O, Tajer C, de Barros E Silva PGM, Roettig ML, Huo Y, Granger CB; IMPACT-AF investigators. A multifaceted intervention to improve treatment with oral anticoagulants in atrial fibrillation (IMPACT-AF): an international, cluster-randomised trial. Lancet. 2017 Oct 14;390(10104):1737-1746. doi: 10.1016/S0140-6736(17)32165-7. Epub 2017 Aug 28. PMID 28859942
- [Derived] Rao MP, Ciobanu AO, Lopes RD, Fox KA, Xian Y, Pokorney SD, Al-Khalidi HR, Jiang J, Kamath DY, Berwanger O, Xavier D, Bahit CM, Tajer C, Vinereanu D, Huo Y, Granger CB. A clustered randomized trial to IMProve treatment with AntiCoagulanTs in patients with Atrial Fibrillation (IMPACT-AF): design and rationale. Am Heart J. 2016 Jun;176:107-13. doi: 10.1016/j.ahj.2016.03.011. Epub 2016 Mar 21. PMID 27264227